CLINICAL TRIAL: NCT07107269
Title: Diet and Microbiome Interactions: Application in Posttraumatic Stress Disorder
Brief Title: Diet and Microbiome Interactions: Application in Posttraumatic Stress Disorder in Adults Consuming Vegetable Drinks
Acronym: DMAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Tiffany Weir, Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 5886
Record Dates: First submitted 2025-07-23; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; Post Traumatic Stress Disorder; Highly Diverse Fruit and Vegetable Drink; PTSD and microbiome
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, parallel arm, controlled diet intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High plant diversity intervention (Experimental): 30 different vegetables as a 4 oz blended beverage in a mylar pouch.
  Interventions: Other: Functional Food intervention
- Low plant diversity intervention group (Experimental): 3 vegetable blend as a 4 oz blended beverage in a mylar pouch.
  Interventions: Other: Low plant diversity beverage

INTERVENTIONS:
Other: Low plant diversity beverage — Blended drink made from 3 organic vegetables (Power Greens mix)
  Arms: Low plant diversity intervention group
Other: Functional Food intervention — This is a 4oz shot made from 30 different organic vegetables and packaged in mylar pouches.
  Arms: High plant diversity intervention

SUMMARY:
The gut microbiome has been shown to impact various facets of human health, including mental health. Studies have shown that populations with more agrarian lifestyles tend to have fewer chronic diseases and mental health issues than industrialized populations. A possible factor in these differences is the loss of co-evolved gut microbial taxa that has occurred with Westernization. This hypothesis, termed "Old Friends Hypothesis" suggests that the loss of certain gut microbes leads to immune dysregulation and increased chronic inflammation that contributes to development of cancers, cardiometabolic diseases and even neuroinflammation that can lead to negative behavioral and mental health outcomes. Other studies have shown that increasing the intake of plant foods may help increase diversity of the microbes in the gut and that this increased diversity could lead to better health outcomes in humans.

The investigators propose to evaluate daily consumption of a drink consisting of a high diversity of plants (30 plant species) for four weeks on the diversity of the gut microbiome, biological signatures of inflammation, quality of life, sleep quality, and PTSD symptoms among persons with a diagnosis of PTSD.

The investigators hypothesize that four weeks of daily consumption of this high plant diversity beverage (30 plant species) will increase gut microbiome ɑ-diversity, reduce markers of systemic inflammation, and improve PTSD symptom severity relative to daily consumption of a beverage containing only three plant species.

DETAILED DESCRIPTION:
The intervention will be a double-blind parallel arm study that consists of a four-week treatment period where participants will be randomized to either the experimental or control arm of the study.

During this four-week treatment period the participants will consume either a 4 oz beverage consisting of 30 different blended vegetables (high diversity treatment) or a similar control beverage consisting of 4 oz of blended Power Greens mix, containing only 3 different plant species (low diversity F&V treatment).

The participants will be asked to provide 2-day diet records every two weeks throughout the study. Participants will also complete daily bowel movement records using the Bristol Stool Scale (BSS) and collect 3 fecal samples (baseline, mid-point and final) that will be returned to the clinic at scheduled visits. Blood samples and gut, sleep, and mental health questionnaire data will be collected at the beginning and end of the study.

Primary objectives are as follows:

Objective 1: To determine whether consuming a higher number of plant types, thereby increasing exposure to diverse plant-associated microbes, increases gut microbial diversity. Specifically, investigators will use fecal samples from individuals before and after 4-week consumption of a 4 oz beverage made with high (30 different plants) and low botanical diversity (3 different plants) to assess taxonomic richness (CHAO) and diversity (Shannon) using 16s rRNA and metagenomic sequencing approaches.

Objective 2: To determine how differences in plant diversity consumption influence inflammation and immune signatures, specifically plasma hsCRP levels and number/type of circulating T-regulatory cells. hsCRP will be assayed using ELISA and T-cells and other immune cells will be profiled from collected peripheral blood mononucleocytes (PBMCs) via flow cytometry.

Objective 3: To determine whether gut microbial diversity and inflammatory profiles correlate with PTSD symptom severity. PTSD symptoms will be evaluated at each visit using the PCL-5 assessment and changes with treatment as well as correlates with other primary outcome measures will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (age 18-65) with a diagnosis of PTSD and a BMI <35. Participants should be willing to follow the study protocols and attend all clinic visits.

Exclusion Criteria:

* Exclusion criteria include antibiotic use within the previous three months, BMI>35, vegan or vegetarian diet, allergies to any of the foods included in the intervention beverages, an unstable medication regimen, and diagnosis of diseases such as gastrointestinal diseases, cancer, CVD, diabetes or autoimmune disease and pregnancy or breastfeeding. Specific medication use (other than antibiotics) would not disqualify an individual if they have had a stable medication regimen for at least two months prior to beginning the study and remain on their medication for the study duration. However, medication changes or antibiotic use during the study would be a reason for dismissal Additionally, inclusion or exclusion in the study will be determined case-by-case based on self-reported supplement use or if the individual feels they are unable to adhere to the study requirements, which includes consuming beverages daily, providing stool or blood samples, tracking bowel movements and symptoms, and attending scheduled clinic visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes in self-assessed severity of post-traumatic stress disorder (PTSD) symptoms | From enrollment to the end of the 4-week intervention period.
  PTSD Checklist for DSM-5 or the PCL-5 questionnaire.
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including:
  Monitoring symptom change during and after treatment Screening individuals for PTSD Making a provisional PTSD diagnosis
  A higher score on the PCL-5 indicates a greater level of distress and impairment associated with PTSD symptoms. The total score ranges from 0 to 80, with higher scores reflecting a more severe symptomatology. A total score of 32 or above suggests the presence of clinically significant PTSD symptoms, which may require further assessment and treatment.
Gut Microbiota Richness | From enrollment to the end of the 4-week intervention period.
  Microbiota richness will be determined by the number of amplicon sequence variants (actual or estimated) in a fecal sample.
Gut microbiota diversity | From enrollment to the end of the 4-week intervention period.
  The Shannon-Wiener index will be applied to 16s rRNA amplicon sequence variants to determine microbial community diversity within a fecal sample.
C-reactive protein in plasma | From enrollment to the end of the 4-week intervention period.
  CRP, or C-reactive protein, is a substance produced by the liver in response to inflammation in the body. It is commonly measured in blood using a high sensitivity ELISA test to assess general inflammation levels, helping to identify underlying health issues such as infections, tissue injury, or chronic inflammatory diseases. Elevated levels of CRP are associated with PTSD.

SECONDARY OUTCOMES:
Seated Blood Pressure | From enrollment to the end of the 4-week intervention period.
  Average of 3 seated brachial blood pressure readings taken in the clinic at each visit.
Changes in T-cell populations | From enrollment to the end of the 4-week intervention period.
  Using flow cytometry to look at the number and types of T-cells in peripheral blood mononuclear cells can be used to look at changes in immune response and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Weir, PhD, Principal Investigator — Colorado State University
Locations (1):
- Food and Nutrition Clinical Research Lab - Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No